CLINICAL TRIAL: NCT03309189
Title: National Studie Gesundheit Und Ernährung Von Primarschülern
Brief Title: Swiss Childhood Health and Nutrition Survey
Acronym: CHildHNS
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Senior Scientist, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: CHildHNS
Record Dates: First submitted 2017-08-18; First posted 2017-10-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Overweight and Obesity in Schoolchildren
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to assess the prevalence of overweight and obesity in 6 to 12 year old children in Switzerland. This data will be used to investigate trends in the development of overweight and obesity in Switzerland. In addition, a questionnaire will be used to assess data on physical activity, nutrition, health and socioeconomic background and waist circumference as well as skin fold thicknesses will be measured.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 12 years

Exclusion Criteria:

* none

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children at the selected schools and in the defined age range are eligible.
Sampling Method: Probability Sample
Enrollment: 2292 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of overweight and obesity | 1 day of first visit
  Based on weight and height measurements BMI z-scores will be calculated for the classification in the different weight status groups (underweight, normal weight, overweight, obese)

SECONDARY OUTCOMES:
Waist circumference | 1 day of first visit
body fat % | 1 day of first visit
  Based on the measurement of skinfold thicknesses at 4 sites body fat % will be calculated
Physical activity | 1 day of first visit
  Assessed using a questionnaire
Nutrition | 1 day of first visit
  Assessed using a questionnaire
General health | 1 day of first visit
  Assessed using a questionnaire
Socioeconomic background | 1 day of first visit
  Assessed using a questionnaire

OTHER OUTCOMES:
Age | 1 day of first visit
  Assessed using a questionnaire
Gender | 1 day of first visit
  Assessed using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No